CLINICAL TRIAL: NCT02309853
Title: Visual and Tactile Scanning Training in Patients With Neglect After Stroke
Acronym: ViTaTrain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HES-SO Valais-Wallis (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P40907
Record Dates: First submitted 2014-11-09; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Hemispatial Neglect
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual and tactile scanning training (Experimental): 20 Sessions of 30 minutes with a visual and tactile scanning training in the personal, peripersonal and extrapersonal space combined with trunk rotation
  Interventions: Other: Visual and tactile scanning training
- Unimodal visual scanning training (Active Comparator): 20 sessions of 30 minutes with traditional uni-modal visual scanning training
  Interventions: Other: Uni-modal visual scanning training

INTERVENTIONS:
Other: Visual and tactile scanning training — 20 Sessions of 30 minutes with a visual and tactile scanning training in the personal, peripersonal and extrapersonal space and trunk rotation. The intervention includes visual or tactile scanning training in three different spaces and will be individually adapted to the needs of the patients.
  1. Visual or tactile scanning in the personal space
  2. Visual or tactile scanning and trunk rotation in the peripersonal space
  3. Visual scanning and trunk rotation in the extrapersonal space
  Arms: Visual and tactile scanning training
Other: Uni-modal visual scanning training — 20 sessions of 30 minutes with traditional uni-modal visual scanning training in the peripersonal space.
  Arms: Unimodal visual scanning training

SUMMARY:
The purpose of this study is to evaluate whether 20 Sessions of 30 minutes with a visual and tactile scanning training in the personal, peripersonal and extrapersonal space combined with trunk rotation will be feasible and provide better results compared to 20 Sessions of 30 minutes of a standard visual scanning programme.

DETAILED DESCRIPTION:
In patients with stroke, unilateral neglect is a predictor for poor independency and quality of life. Current therapies are lacking a progression of intensity based on clear criteria. In addition, therapies include rather analytical exercises and the transfer of the achieved functions to activities of daily living remains difficult. Therefore, the investigators developed a criterion based system, in which the investigators are matching interventions to specific neglect related deficits and behaviour. The investigators plan a randomised controlled trial (stage 2 "development of concept trial") to evaluate whether an Experimental Group with 20 Sessions of 30 minutes with a visual and tactile scanning training in the personal, peripersonal and extrapersonal space combined with trunk rotation or a Control Group with 20 Sessions of 30 minutes of a standard visual scanning programme results in larger improvements on the neglect behaviour during activities of daily life (Catherine Bergego Scale). Sixteen stroke patients with left side neglect (i.e. right brain lesions) will be recruited in an inpatient rehabilitations setting.

ELIGIBILITY:
Inclusion Criteria:

* First or second time right hemispheric stroke (haemorrhagic or ischaemic, diagnosed with computer tomography or magnetic resonance imaging)
* Time after last stroke: less than 8 weeks
* Hemispatial neglect with at least seven points on the Catherine Bergego Scale
* Right handed

Exclusion Criteria:

* Reduced vision after rectification (i.e. corrected vision sufficient to read newspaper-sized print)
* Mini-Mental State Evaluation Score below 11
* Not fluently speaking and understanding French or German language in order to understand the tasks and the assessments, as assessed and judged by the medical doctor and the staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Neglect behaviour during activities of daily life measured with the Catherine Bergego Scale | up to 14 months
  Measured with the Catherine Bergego Scale
Adherence rate of the patients to the treatment | up to 11 months

SECONDARY OUTCOMES:
Visual neglect measured with the Behavioural Inattention Test (conventional subtest) | up to 14 months
  Measured with the Behavioural Inattention Test (conventional subtest)
Severity of disability in a rehabilitation setting measured with the Functional Independence Measure | up to 11 months
  Measured with the Functional Independence Measure
Personal neglect measured with the Vest Test | up to 14 months
  Measured with the Vest Test
Mobility related disability easured with the Rivermead Mobility Index | up to 11 months
  Measured with the Rivermead Mobility Index
Health related quality of life measured with the EQ-5D | up to 14 months
  Measured with the EQ-5D
Length of stay in inpatient rehabilitation setting | up to 11 months
Inclusion rate and refusal rate per week | up to 11 months
Completeness of documents | up to 11 months
Length of time of assessments | up to 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sattelmayer, MSc, MA, Principal Investigator — HES-SO Valais-Wallis
Locations (1):
- Berner Klinik Montana, Montana, Valais, Switzerland